CLINICAL TRIAL: NCT01615965
Title: Detection of Micrometastases in Lymph Nodes of Patients With Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2607/09
Record Dates: First submitted 2010-02-27; First posted 2012-06-11 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; lymph node; micrometastasis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Micrometastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- micrometastases (Experimental): Molecular biologic detection of micrometastases in lymph nodes of patients with localized prostate cancer treated with radical prostatectomy and lymphadenectomy.
  Interventions: Other: tumor marker detection in lymph nodes

INTERVENTIONS:
Other: tumor marker detection in lymph nodes — tumor marker detection in lymph nodes by quantitative PCR

SUMMARY:
The purpose of this study is to set up a model for detecting micrometastases in Lymph nodes of patients with prostate cancer by quantitative polymerase chain reaction and its impact on progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate cancer
* Locally operable tumor
* Negative bone scan (obligatory if Gleason Score > 7 or PSA > 20ng/ml
* Karnofsky ≥ 80%
* Age 18 - 75 years
* Informed consent in written form
* Sufficient hematologic, coagulatory and renal function
* Compliant patient and geographic precondition for adequate follow-up given

Exclusion Criteria:

* Manifest secondary tumor
* Organ metastases on CT-scan /MRI or in Histology
* Myocardial infarction or stroke within the last 6 months
* Severe cardiovascular (Grade III - IV according to NYHA), pulmonary (pO2 < 60 mmHg), renal, hepatic oder hematopoetic impairment
* Severe active or chronic infection (z.B. pos. HIV-Antibody-Test, HBs-Ag-detected in Serum and/ or chronic Hepatitis)
* Severe psychiatric disease
* Previous chemotherapy
* Previous pelvine radiotherapy

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-02; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical recurrence free survival | 2 years
  Influence of molecularbiologic micrometastases in lymph nodes on biochemical recurrence free survival in comparison with patients who have histopathologic macrometastases or no evidence of lymph node metastases

SECONDARY OUTCOMES:
Frequency of molecular detected lymph node micrometastases according to their topography | 2 years
  Description of the anatomic distribution of molecularbiologic lymph node micrometastases in prostate cancer patients treated with radical prostatectomy and extended lymphadenectomy.
  The frequency of molecular detected lymph node micrometastases according to their anatomic distribution at the obturatoric fossa, external iliac, internal iliac and common iliac arteries´ region will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Urologic Department, Munich, Germany

REFERENCES:
- See also: Related Info — http://www.mriu.de